CLINICAL TRIAL: NCT04169932
Title: The Clinical Study of CD20 CAR-T Cells in Patients With Relapsed and Refractory B Cell Non-Hodgkin Lymphoma
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Longyao Biotechnology Inc., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20191023V1.1
Record Dates: First submitted 2019-11-08; First posted 2019-11-20 (Actual); Last update posted 2019-11-20 (Actual); Status verified 2019-11

CONDITIONS: Relapsed and Refractory B Cell Lymphoma; Non-Hodgkin Lymphoma
Keywords: CD20 CAR T Cells; Safety, tolerance and efficacy
MeSH Terms: conditions — Recurrence; Lymphoma, B-Cell; Lymphoma, Non-Hodgkin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CD20 CAR-T (Experimental)
  Interventions: Biological: CD20 CAR-T

INTERVENTIONS:
Biological: CD20 CAR-T — The maximum dose was determined according to the dose escalation test. Based on the number of CART cells per kg body weight which was proved to be safe and effective, all the subjects were treated with one single dose of CD20 CART cells per treatment course. The dose escalation test was designed to evaluate the four dose levels of CD20-CART (1 × 10 ^ 6 cells/kg,2 × 10 ^ 6 cells/kg,4 × 10 ^ 6 cells/kg,8 × 10 ^ 6 cells/kg).

SUMMARY:
This is a single arm, open-label study to evaluate the safety, tolerance and efficacy of CD20 CAR-T Cells in patients with relapsed and refractory B cell non-Hodgkin Lymphoma. Subjects receive a single intravenous infusion of CD20-CART cells per treatment course.

DETAILED DESCRIPTION:
The maximum dose was determined according to the dose escalation test. Based on the number of CART cells per kg body weight which was proved to be safe and effective, all the subjects were treated with one single dose of CD20 CART cells per treatment course. The dose escalation test was designed to evaluate the four dose levels of CD20-CART (1 × 10 ^ 6 cells/kg,2 × 10 ^ 6 cells/kg,4 × 10 ^ 6 cells/kg,8 × 10 ^ 6 cells/kg). Each CD20-CART infusion will be carried out on day 0. Each subject was observed for at least 4 weeks after the last infusion. If there was no dose-limited toxicity (DLT), it is necessary to continue multiple treatment courses at this dose level. The detailed administration time and dose were decided by the researchers. The observation period was 4 weeks after the end of the course of treatment. If 2 or more cases of DLT occurred at a certain dose level, the prior dose level was the maximum tolerable dose of (MTD). If one case of DLT occurred, 3 subjects were added to the group. If there were no DLT in 3 cases, the next dose level would be estimated. If at least 1 case of DLT occurred in the 3 cases, the prior dose was the maximum tolerated dose of (MTD). If there were no DLT at the maximum dose, the maximum tolerant dose was the maximum dose.

ELIGIBILITY:
Inclusion Criteria:

* 1. Patients with CD20+ relapsed or refractory B cell Non-Hodgkin lymphoma, which includes but not limited to diffuse large B cell lymphoma (DLBCL), follicular lymphoma, transformed follicular lymphoma, marginal-zone lymphoma, mantle-cell lymphoma, small B-cell lymphoma, are eligible for inclusion in this study must meet one of the following criteria:

  1. Relapsed or refractory as defined by not achieving a PR after a second-line drug therapy such as CD20 monoclonal antibodies, or achieving a PR but the disease has progressed, or chieving a CR but the disease has relapsed.
  2. Relapse after autologous stem cell transplantation (SCT) within 1 year.
* 2. Adult subjects between 18 and 70 years of age, inclusive.
* 3. Life expectancy > 3 months.
* 4. ECOG score between 0 and 1.
* 5. Liver, Renal, Heart and Lungs function defined as:

  1. Creatininec≤1.5 ULN;
  2. ALT/AST ≤2.5 ULN;
  3. Total Bilirubin≤1.5×ULN;
  4. Pulse oxygenation≥92%;
  5. Left Ventricular Shortening Fraction (LVSF)≥50%;
  6. Echocardiogram (ECHO) shows no obvious pericardial effusion.
* 6. According to Lugano 2014 criteria for assessing FDG-PET/CT in lymphoma, the lesions must meet the minimum size requirement of being >15 mm in longest diameter (LDi).
* 7. Subjects could comprehend the clinical study and able to provide written consent at the time of consent or assent.

Exclusion Criteria:

* 1. Pregnant or lactating women, or women with pregnancy plans within 6 months.
* 2. HBsAg or the titer of HBV was not in the range of normal reference value; positive for presence of HCV antibody or HCV RNA in peripheral blood; positive for presence of human immunodeficiency virus type 1 or 2 (HIV-1 or HIV-2).
* 3. Severe heart disease: include but not limited to Unstable angina pectoris, myocardial infarction (within 6 months before screening), Congestive heart failure (New York Heart Association [NYHA] Classification ≥ III).
* 4. Previously received other CART therapy or transgenic cell therapy.
* 5. The subjects participated in clinical trials within 6 months before screening.
* 6. Subjects who were receiving systemic steroid therapy and determined by the researchers to require long-term use of systemic steroid therapy except for inhalation or local use before screening.
* 7. Subjects who had more than 2 years of autoimmune disease history (such as Crohn's disease, rheumatoid arthritis, systemic lupus erythematosus) that caused organ damage or subjects who needed to take systemic immunosuppressants;
* 8. Any unstable systemic disease, including but not limited to, liver, kidney or metabolic diseases requiring drug treatment.
* 9. Autologous transplantation or allotransplantation was performed within 6 months after admission.
* 10. Evidence or history of central nervous system involvement in lymphoma.
* 11. Subjects with active bleeding caused by the involvement of the original lesion in the digestive tract.
* 12. Subjects with active infectious diseases who received systematic antibiotic treatment within 2 weeks of admission.
* 13. Other subjects judged by the researchers to be unsuitable for admission to the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-11-22 (Estimated); Primary Completion 2022-11-22 (Estimated); Study Completion 2022-11-22 (Estimated)

PRIMARY OUTCOMES:
The Adverse events (AEs) | 4 weeks
  Number of Participants With Treatment-Related Adverse Events as Assessed by CTCAE v4.0
Expression of CD20 CART cells | 2 years
  Expression of CD20 CART cells detected by flow cytometry in blood and bone marrow
Detection of CD20 CART cells | 2 years
  Detection of CD20 CART cells in blood, bone marrow by Quantitative Polymerase Chain Reaction (q-PCR).
Graft Activity Endpoint Detection | 2 years
  The vector copy number (VCN) of the exogenous CAR vector in the blood and bone marrow.

SECONDARY OUTCOMES:
Overall remission rate (ORR) | 2 years
Complete Remission (CR) | 2 years
Partial Remission (PR) | 2 years
To evaluate the duration of remission (DOR) | 2 years
To evaluate the Progression-free survival (PFS) | 2 years
To evaluate the Overall survival (OS) | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Yi Yao, ph.D, Study Chair — Shanghai Longyao Bio-Tech Co., Ltd.
Locations (1):
- The First Affiliated Hospital with Nanjing Medical University, Nanjing, Jiangsu, China